CLINICAL TRIAL: NCT03268304
Title: Feasibility of Two Novel Interactive Software Modules for the Rehabilitation of Patients With Neuromuscular Upper Limb Impairments Using the YouGrabber Training System - the KAYO Study Protocol
Brief Title: Feasibility of Two New Software Modules for the Rehabilitation of Patients With Neuromuscular Upper Limb Impairments
Status: Withdrawn | Type: Observational
Why Stopped: The software modules were not completed.
Sponsor: Reha Rheinfelden (Other)
Responsible Party: Principal Investigator, Frank Behrendt, Principal Investigator, Reha Rheinfelden
Other Study IDs: KAYO
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Stroke; Parkinson Disease; Traumatic Brain Injury; Guillain-Barre Syndrome
Keywords: Upper Limb Motor Function Deficit; Neurorehabilitation; Virtual Reality; Action Research Arm Test
MeSH Terms: conditions — Stroke; Parkinson Disease; Brain Injuries, Traumatic; Guillain-Barre Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: VR-based training including AO and MI — Virtual Reality-based training intervention including Action Observation and Motor Imagery using the YouGrabber® training device

SUMMARY:
Introduction: In the recent past, medical training systems using virtual reality (VR) have been introduced to neurorehabilitation to train motor function deficits in patients. The usage of VR-based training systems is based on the evidence of neuroplasticity, which is responsible for recovery of patients suffering from motor dysfunction. Such systems are increasingly used to encourage purposeful limb movements in a VR environment and its efficacy has been found comparable with conventional therapeutic intervention. VR training systems, e.g. the YouGrabber® (YG), will increasingly also be used at home. Therefore, it is essential to integrate valid and reliable assessment tools to monitor the recovery process.

Objectives: The aim of the clinical study is to evaluate the usability, feasibility and validity of the digital version of the ActionResearchArmTest (d-ARAT) using the YG system as a platform. Additionally, the feasibility and usability of the implementation of two rehabilitation measures that only recently became integral part of neurorehabilitation, e.g. Action Observation (AO) and Motor Imagery (MI), into the YG training software will be evaluated. Patients & methods: This observational study is designed as a single-arm trial for testing the assessment software including pre- to post rehabilitation comparison of a training involving AO and MI. Therefore, 75 adult patients with Parkinson's disease, MS, Stroke, traumatic brain injury or Guillain-Barré syndrome will be included. 30 out of the 75 patients will take part in the 4-week training on the enhanced VR-based system with a total of 16 training sessions of 45 min each. Primary outcomes will be the score on the System Usability Scale (SUS) and the ARAT as well as the d-ARAT scores. Secondary outcomes will be hand dexterity (Box-and-Block Test), upper limb activities of daily living (CAHAI) and quality of life (EQ-5D-5L).

Hypothesis: The study was designed to evaluate the d-ARAT and the training software modules for the YG system. Currently AO and MI specific tasks are being integrated and the ARAT subscales will be implemented on the basis of the redesigned glove equipped with new sensors. The results are expected to give recommendations for necessary modifications. They might also contribute knowledge concerning the application of AO and MI tasks within VR training.

ELIGIBILITY:
Inclusion Criteria:

* Patients with motor function impairments of one or both upper limbs caused by Parkinson's disease, MS, Stroke, traumatic brain injury or Guillain-Barré syndrome
* Able to sit in a normal chair without armrests
* Able to score at least one in the Box and Block Test (BBT)
* Comprehend German
* Informed Consent as documented by signature

Exclusion Criteria:

* Wrist-, hand- or finger contractures or an unconsolidated upper limb fracture
* Severe cognitive deficits: Mini-Mental-Status-Test (MMSE) ≤ 20
* Severe spatial-visual disorders, e.g. severe visual neglect
* History of epileptic seizures triggered by visual stimuli (e.g. television, video games) within the last six months
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Full score in the Chedoke Arm and Hand Activity Inventory (CAHAI) assessment
* Brain pacemaker

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. Patients will be recruited from the clinics' inpatient or outpatient departments by physicians, therapists and nurses.
  2. Patients will be recruited from the clinics' patient database. Datasets will be screened for study selection criteria by the involved study personnel. If patients are eligible, they will be sent a letter describing the study and including patient information. If patients are interested in participating, they can contact the study personnel in the clinic by phone or email.
  3. Patients will be recruited via a study information flyer provided on the clinic's homepage and through patient self-help groups. If patients are interested in participating, they can contact the study personnel in the responsible clinic by phone or email.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
cARAT | 17 weeks
  Score on the conventional Action Research Arm Test
dARAT | 17 weeks
  score on the digital ARAT
SUS | 15 weeks
  System Usability Scale questionnaire

SECONDARY OUTCOMES:
BBT | 17 weeks
  Box and Block Test
CAHAI | 17 weeks
  Chedoke McMaster Arm and Hand Activity Inventory
EQ-5D-5L | 17 weeks
  EuroQol five dimensions questionnaire with five-level scale
PGIC | 11 weeks
  Patient Global Impression of change

CONTACTS AND LOCATIONS:
Overall Officials: Frank Behrendt, PhD, Principal Investigator — Reha Rheinfelden; Corina Schuster, PhD, Principal Investigator — Reha Rheinfelden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Behrendt F, Schuster-Amft C. Using an interactive virtual environment to integrate a digital Action Research Arm Test, motor imagery and action observation to assess and improve upper limb motor function in patients with neuromuscular impairments: a usability and feasibility study protocol. BMJ Open. 2018 Jul 16;8(7):e019646. doi: 10.1136/bmjopen-2017-019646. PMID 30012780